CLINICAL TRIAL: NCT06187883
Title: Does Obesity EffectThe Successful Response to the Pulsed Radiofrequency of Lateral Femoral Cutaneous Nerve in Meralgia Parestetica? : A Retrospective Cohort Study
Brief Title: Pulsed Radiofrequency of Lateral Femoral Cutaneous Nerve
Status: Completed | Type: Observational
Sponsor: Mersin Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Suna Aşkın Turan, Pain Department Physician, Mersin Training and Research Hospital
Other Study IDs: MersinTRHlfcn
Record Dates: First submitted 2023-12-06; First posted 2024-01-03 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Meralgia Paresthetica
Keywords: meralgia parestetica; pulsed radiofrequency; obesity; dn4; neuropathic pain
MeSH Terms: conditions — Femoral Neuropathy; Obesity; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: patients treated with PRFT

SUMMARY:
In the current retrospective cohort study, conducted by both pain specialists and neurophysiologists, the primary outcome was to search for the effect of obesity on the efficacy of PRF of LFCN in refractory MP for 6 months. Secondary outcomes were to identify the clinical and diagnostic features of the MP.

DETAILED DESCRIPTION:
In the current retrospective cohort study, conducted by both pain specialists and neurophysiologists, the primary outcome was to search for the effect of obesity on the efficacy of PRF of LFCN in refractory MP for 6 months. Secondary outcomes were to identify the clinical and diagnostic features of the MP.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years treated with PRF neuromodulation of LFCN for MP
* followed up at least 6 months in the pain clinic of the tertiary hospital between January 2020 and August 2023.

Exclusion Criteria:

* inadequate follow-up or missing documentation
* If a new analgesic drug was prescribed during the follow-up period that could affect the evaluation of outcomes, the patients were also excluded.
* Patients who missed appointments, or were unable to communicate with; were not included in the study.
* Patients with secondary entrapment neuropathy (e.g., diabetes, inflammatory arthritis, hypothyroidism), malignancy, pregnancy, skin infection in the inguinal region or dermatitis, lumbar radiculopathy, polyneuropathy, and cardiac pacemakers were excluded.
* In the SSEP analysis, when the latency of LFCN was not evaluated in both sides, these patients were not also included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients older than 18 years treated with PRF neuromodulation of LFCN for MP and followed up at least 6 months in the pain clinic of the tertiary hospital between January 2020 and August 2023.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
response to PRF | 6 months
  loss of neuropathic pain, lasting at least 6 months was defined as a positive categorical outcome. Neuropathic pain was assessed with Douleur Neuropathique 4 questionnaire (DN4) at baseline, and at 1., 3, 6 months by the pain specialist authors. DN4 consisted of 10 items. The first seven items were associated with the patients' subjective compliants related to pain and sensational variations while the last three items were associated with the clinical findings. Those patients who had a score ≥ 4were considered to have neuropathic pain. Patients with a positive outcome at the 1 or 3 month follow-up,but did not come again were excluded from the study. After the data collection, the patients wer divided into two groups: responders with a positive outcome and nonresponders with a negative outcome.MP for 6 months. Age, sex, body mass index (BMI), employment, tight clothing, belts, carrying things at the back of pants were asked in detail at the initial visit of the Pain Clinic.

SECONDARY OUTCOMES:
Secondary outcomes were to identify the clinical and diagnostic features of the MP | 6 months
  Secondary outcomes were to identify the clinical and diagnostic features of the MP. The outcome was assesed by the clinical and electrophysiological data collected from the hospital records. The data was analyzed deeply.

CONTACTS AND LOCATIONS:
Overall Officials: Aşkın Turan, MD, Study Chair — Mersin Şehir Hastanesi
Locations (1):
- Suna Aşkın Turan, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The Data and materials are available from the corresponding author upon reasonable request and are subject to ethical review.